CLINICAL TRIAL: NCT00989872
Title: A Randomized, Double-blind, Placebo-Controlled, Ascending Single-Dose Safety, Tolerability, and Pharmacokinetics Study of EDP-322 in Healthy Adult Volunteers
Brief Title: Safety and Pharmacokinetics of Ascending Single Oral Doses of EDP-322 in Nonfasting and Fasting Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Responsible Party: Maria T. Madison, Dir. Clinical Operations, Enanta Pharmaceuticals
Allocation: Randomized | Masking: Triple | Purpose: Treatment
Other Study IDs: EDP-322-007-001
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Last update posted 2009-10-06 (Estimated); Status verified 2009-10

CONDITIONS: Skin and Soft Tissue Infections; Methicillin-resistant Staphylococcus Aureus
Keywords: Macrolides; Antibiotics; Safety; Tolerability; Pharmacokinetics; Phase I; MRSA/SSTI
MeSH Terms: conditions — Soft Tissue Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: EDP-322

SUMMARY:
This was a randomized, double-blind, placebo-controlled, ascending single dose safety, tolerability, and pharmacokinetic study of orally administered EDP-322. This study was conducted at a single site. EDP-322 has a benefit to risk profile that supports testing in target patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males or females [if documentation existed that they were surgically sterilized].
* Were in good general health as determined by medical history, physical exam and clinical laboratory tests, and without evidence of clinically significant abnormality, in the opinion of the Investigator and Medical Monitor.
* The resting 12-lead ECG obtained at Screening shows no clinically significant abnormality and a QTc (Bazett's correction) <450 msec.
* Weight less than 132 pounds (60kg) with BMI between 18-32 kg/m3, inclusive.
* Subject has read, understood, and signed the written informed consent form.

Exclusion Criteria:

* History of chronic or recurrent renal, hepatic, pulmonary, allergic, cardiovascular, gastrointestinal, endocrine, central nervous system, hematologic or metabolic diseases, or immunologic, emotional and/or psychiatric disturbances.
* History of gastric surgery, vagotomy, bowel resection, or any surgical procedure that might interfere with gastrointestinal motility, pH, or absorption.
* Any abnormal or screening clinical lab test results...
* Medication Related exclusions...
* Lifestyle related...

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)

PRIMARY OUTCOMES:
The study objectives included determining the safety, tolerability and pharmacokinetics of single oral doses of EDP-322 in healthy adult volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L Hunt, MD, PhD, Principal Investigator — PPD Phase I Unit
Locations (1):
- PPD Phase I Unit, Austin, Texas, United States